CLINICAL TRIAL: NCT00473200
Title: Effect of Oral S-adenosylmethionine (SAMe) on Blood Levels of Homocysteine in Human Subjects
Brief Title: Effect of S-adenosylmethionine (SAMe) on Blood Levels of Homocysteine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 005-210
Record Dates: First submitted 2007-05-10; First posted 2007-05-14 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Hyperhomocysteinemia
Keywords: hyperhomocysteinemia; homocysteine; S-adenosylmethionine; SAMe; Asymmetric dimethylagrinine (ADMA)
MeSH Terms: conditions — Hyperhomocysteinemia | interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S-adenosylmethionine (Active Comparator): S-adenosylmethionine
  Interventions: Dietary Supplement: S-adenosylmethionine
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: S-adenosylmethionine

INTERVENTIONS:
Dietary Supplement: S-adenosylmethionine — 1200 mg daily

SUMMARY:
The purpose of this study is to investigate whether S-adenosylmethionine (SAMe), a natural substance available as a nutritional supplement, can influence blood levels of homocysteine (Hcy). More specifically, we will determine if chronic oral SAMe administration affects homocysteine metabolism in patients with vascular disease who have mild to moderate hyperhomocysteinemia.

DETAILED DESCRIPTION:
The purpose of this study is to investigate whether S-adenosylmethionine (SAMe), a natural substance available as a nutritional supplement, can influence blood levels of homocysteine (Hcy). More specifically, we will determine if chronic oral SAMe administration effects homocysteine metabolism in patients with vascular disease who have mild to moderate hyperhomocysteinemia through the following specific aims:

Specific Aim 1 - To determine the effect of oral SAMe (1200 mg/day) on plasma total homocysteine levels in subjects with mild to moderate hyperhomocysteinemia.

Specific Aim 2 - To determine the effect of oral SAMe (1200 mg/day) with and without supplementation of folate, vitamin B12 and B6, on plasma homocysteine levels in patients with mild to moderate hyperhomocysteinemia.

Specific Aim 3 - To determine the effect of oral SAMe (1200 mg/day) on plasma levels pf asymmetric dimethylarginine (ADMA) in subjects with mild to moderate hyperhomocysteinemia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Must have a serum homocysteine value greater than or equal to 14 μmol/L
* Stable weight 3 months prior to study participation

Exclusion Criteria:

* Subjects with a BMI greater than 35 or less than 18
* Currently taking B 100 or other high-dose B vitamin supplements within the past 12 months
* Taken methionine or SAMe supplements within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To determine the effect of oral SAMe (1200 mg/day) on plasma total homocysteine (tHcy) and asymmetric dimethylagrinine (ADMA) levels in subjects with mild to moderate hyperhomocysteinemia. | 6 weeks

SECONDARY OUTCOMES:
To determine the effect of oral SAMe (1200 mg/day) with and without supplementation of folate, vitamin B12 and B6, on plasma homocysteine levels in patients with mild to moderate hyperhomocysteinemia. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teodoro Bottiglieri, PhD, Study Director — Baylor Research Institute
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States